CLINICAL TRIAL: NCT02103504
Title: Roentgen Stereophotogrammetric Analysis (RSA) of the ATTUNETM Posterior Stabilized Fixed Bearing Knee System
Brief Title: DePuy Attune Total Knee Arthroplasty RSA Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Dunbar (Other)
Collaborators: Concord Hospital (Other); Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor-Investigator, Michael Dunbar, Orthopedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEP ATT
Record Dates: First submitted 2014-03-28; First posted 2014-04-04 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DePuy Attune TKA (Other): DePuy Attune posterior stabilized fixed bearing total knee replacement
  Interventions: Device: DePuy Attune posterior stabilized fixed bearing total knee replacement

INTERVENTIONS:
Device: DePuy Attune posterior stabilized fixed bearing total knee replacement

SUMMARY:
The DePuy Attune knee system incorporates several key features aimed at improving kinematics of the knee joint, range of motion, and smoothness of use compared to existing total knee replacement technologies. As this is a newly approved medical device, clinical testing in patients using high precision diagnostics is important to evaluate the stability of implant fixation and in vivo function. We propose a multi-centre consecutive series study examining the stability of the Attune posterior-stabilized knee design in 30 patients undergoing total knee arthroplasty for a follow-up period of 2 years. Radiostereometric analysis (RSA) will be utilized to identify the micromotion of the tibial tray with respect to the surrounding bone. Health status and functional outcome measures will be recorded to quantify functional status of subjects before surgery and at follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating primary total knee arthroplasty
* Between the ages of 21 and 80 inclusive
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria:

* Active or prior infection
* Medical condition precluding major surgery

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Implant migration | 2 years

SECONDARY OUTCOMES:
Functional range of motion | 2 years
Self-reported health status | 2 years
  EQ-5D score
Self-reported joint status | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunbar, Principal Investigator — Capital Health, Canada
Locations (3):
- Canada (3):
  - Concordia Hospital, Winnipeg, Manitoba
  - Capital District Health Authority, Halifax, Nova Scotia
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec